CLINICAL TRIAL: NCT06261996
Title: Safety and Efficacy of Fospropofol vs Propofol During Invasive Mechanical Ventilation in Anesthesiology Intensive Care Unit: A Preliminary Study
Brief Title: Safety and Efficacy of Fospropofol vs Propofol During Invasive Mechanical Ventilation.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Henan Provincial People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: henanFSH
Record Dates: First submitted 2024-02-08; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Invasive Mechanical Ventilation
Keywords: Fospropofol; Propofol; Invasive mechanical ventilation; sedation
MeSH Terms: interventions — fospropofol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fospropofol group (Active Comparator): Fospropofol is administered to patients after admission to the roomat a pumping rate of 1 mg/kg/h.
  Interventions: Drug: Fospropofol
- Propofol group (Placebo Comparator): Propofol is administered after admission to the room at a pumping rate of 0.5 mg/kg/h.
  Interventions: Drug: Fospropofol

INTERVENTIONS:
Drug: Fospropofol — Fospropofol is administered after admission to the room at a pumping rate of 1 mg/kg/h.
  Other Names: fospropofol disodium

SUMMARY:
The goal of this clinical trial is to compare the safety and efficacy of fospropofol and propofol during sedation in invasively mechanically ventilated patients in the Anesthesia Intensive Care Unit (AICU). Specific objectives include the following:

* Evaluate the sedative effects of fospropofol and propofol in invasively mechanically ventilated patients. Compare the sedative effects of the two medications using relevant clinical indicators and scoring tools, such as the Richmond Agitation-Sedation Scale (RASS).
* Compare the safety of fospropofol and propofol during sedation. Monitor medication-related adverse reactions, such as respiratory depression, hypotension, arrhythmias, headache, injection site pain, and assess the differences in adverse reaction incidence between the two medications.
* Compare the characteristics of recovery from sedation between PPD and propofol. Focus on the time from sedation to emergence from sedation and compare the differences in recovery time between the two medications.

Participants will be sedated with fospropofol or propofol during invasive mechanical ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-65 years old
2. Intubation and mechanical ventilation <12h before enrollment
3. Expected to require continuous invasive ventilation and sedation less than 6h after admission to anesthesia intensive care unit (AICU).
4. Signed informed consent

Exclusion Criteria:

1. parturient, childbirth or lactating mothers
2. acute severe neurological disease or coma
3. chronic renal failure
4. previous mechanical ventilation >12h
5. severe liver dysfunction (Child-Pugh score C)
6. BMI >30kg/m2 (>90kg)
7. dying

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-12 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
The patient's Richmond Agitation-Sedation Scale (RASS) score and the incidence of adverse reactions | Admission to the intensive care unit to 2 hours after weaning off the ventilator.
  The participant's RASS score was assessed by the caregiver and the occurrence of adverse reactions was recorded. Adverse effects include hypotension, bradycardia, tachycardia, agitation, pain at the injection site, nausea and vomiting, edema, fever, anemia, paresthesias, headache, and hypoxemia.

SECONDARY OUTCOMES:
Incidence of adverse reactions during the follow-up period | 2 hours after weaning off the ventilator to 24 hours after leaving the intensive care unit.
  Adverse effects include hypotension, bradycardia, tachycardia, agitation, pain at the injection site, nausea and vomiting, edema, fever, anemia, paresthesias, headache, and hypoxemia.
Extubation time | From admission to the intensive care unit to removal of the endotracheal tube
  The time from admission to the intensive care unit to removal of the endotracheal tube

CONTACTS AND LOCATIONS:
Overall Officials: Jiaqiang Q Zhang, M.D, Study Chair — Henan Provincial People's Hospital